CLINICAL TRIAL: NCT05534607
Title: Natives Engaged in Alzheimers Research - 'Ike Kupuna (Elder Wisdom) Project
Brief Title: Natives Engaged in Alzheimers Research - 'Ike Kupuna
Acronym: NEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 'Ike Kupuna
Record Dates: First submitted 2022-08-12; First posted 2022-09-09 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Mild Cognitive Impairment; Subjective Cognitive Impairment
Keywords: MCI; Alzheimer's disease; Alzheimer's disease and related dementias; Vascular dementia; ADRD; SCI; Native Hawaiian and Pacific Islander; NHPI; Hula; cultural based intervention; behavioral intervention
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Intervention Model Description: The study uses a wait list control design, where the wait-list control group is offered the intervention at the completion of the intervention group's 12-month intervention and assessment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will immediately receive the Ola Mau i ka Hula intervention after randomization for 12 months. The intervention program is 8 months with a 4 month self-monitoring period.
  Interventions: Behavioral: Ola Mau i ka Hula
- Wait-list control group (No Intervention): After baseline data collection, participants randomized to the wait-list control arm will not receive the Ola Mau i ka Hula Program while their counterparts who were randomized to the intervention arm are undergoing the intervention program. Thus, they will not be offered the intervention until after the intervention arm is completed and their 12-month follow-up data collection is completed. They will only receive the educational component of the intervention from us during this 12-month period but they will be instructed to continue with their routine medical care as usual.
  Wait-list control group will be offered the opportunity to receive intervention at the conclusion of 12 month assessment period, regardless of whether they were retained for the full 12 months of data collection.

INTERVENTIONS:
Behavioral: Ola Mau i ka Hula — The first 3 months of the hula-based intervention program was designed and standardized as a culturally-based physical activity (PA) that includes 15 minutes of ADRD education and intervention orientation with 12 weeks of hula lessons.
  These hula lessons consist of two 60-minute classes per week over 12 weeks. Each hula lesson will consist of 8 participants, providing them with the opportunity to engage-in this social support network.
  For the remaining 5 months of the Ola Mau i ka Hula Program, hula lessons led by the kumu hula will be reduced to once a month for 60 min. In addition, the intervention group will meet with a community-peer educator weekly over this 5-month period. Each meeting will be 90 minutes in length with 60 minutes of hula practice following the same format as previous classes, and 30 minutes will cover the PILI Lifestyle Plan curriculum and cultural-based cognitive exercises, alternating weekly.
  Other Names: Ola Mau
  Arms: Intervention group

SUMMARY:
This study will conduct a group randomized trial to test the effects of a hula-based intervention in improving vascular risk factors for ADRD and cognitive complaints and function over 12 months.

DETAILED DESCRIPTION:
This study will conduct a pragmatic group-randomized trial (GRT) with NHPIs aged 50-75 years with at least 1 of 4 modifiable vascular risk factors for ADRD (hypertension, hyperglycemia, obesity, or dyslipidemia) and either SCI or MCI using a wait-list control design to test the effects of the hula-based intervention. The primary outcomes will be vascular risk factors for ADRD and subjective cognitive complaints. Secondary outcomes will include measures of cognitive performance, physical function, and mental health.

ELIGIBILITY:
Inclusion Criteria:

1. self-reported Native Hawaiian or other Pacific Islander ancestry;
2. ages 50+ but not older than 75 (optimal age range for preventing future dementia in people with cognitive impairment, above 75 is not likely to benefit from this study given their advance age);
3. has subjective cognitive impairment (SCI) or mild cognitive impairment (MCI);
4. have a diagnosis of hypertension, diabetes, dyslipidemia, or obesity (body-mass-index ≥ 30 kg/m2);
5. physically able and willing to engage in moderate physical activity necessary for Hula; and
6. physician's approval to participate in moderate physical activity

Exclusion Criteria:

1. currently pregnant;
2. already actively practicing Hula at least once per week; or
3. clinical diagnosis of ADRD (mild to severe); or
4. current diagnosed major depressive disorder at moderate or greater stage, or moderate or greater depression on the Center for Epidemiological Studies Depression Scale (CES-D).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in participants' systolic blood pressure at each time frame from baseline | 3 months, 8 months, 12 months
  Vascular risk factor assessed using Omron©HEM-907XL
Change in participants' Hemoglobin A1c at each time frame from baseline | 12 months
  Vascular risk factor assessed using Alere Cholestech LDX® System
Change in participants' total cholesterol at each time frame from baseline | 3 months, 8 months, 12 months
  Vascular risk factor assessed using Alere Cholestech LDX® System
Change in participants' body mass index at each time frame from baseline | 3 months, 8 months, 12 months
  Vascular risk factor assessed using Tanita BWB800AS scale
Change in participants' Cognitive Change Index score at each time frame from baseline | 3 months, 8 months, 12 months
  Cognitive function assessed using Cognitive Change Index assessment
Change in participants' Number Symbol Coding Test score at each time frame from baseline | 3 months, 8 months, 12 months
  Cognitive function assessed using Number Symbol Coding Test
Change in participants' overall Cognivue score at each time frame from baseline | 3 months, 8 months, 12 months
  Cognitive function assessed using Cognivue device
Change in participants' overall Quick Dementia Rating System score at each time frame from baseline | 3 months, 8 months, 12 months
  Cognitive function assessed using Quick Dementia Rating System assessment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Kaholokula, PhD, Principal Investigator — University of Hawaii
Locations (3):
- United States (3):
  - Kula No Na Po'e, Honolulu, Hawaii
  - Kokua Kalihi Valley, Honolulu, Hawaii
  - Hui No Ke Ola Pono, Wailuku, Hawaii